CLINICAL TRIAL: NCT00907608
Title: A Proof-of-Concept Study of Darbepoetin Alfa in Partial Correction of Anemia in Chinese With Diabetic Nephropathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to difficulty in patient recruitment
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Dr Peter CY Tong, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PWH-2008-darbe
Record Dates: First submitted 2009-05-21; First posted 2009-05-22 (Estimated); Last update posted 2009-05-22 (Estimated); Status verified 2009-05

CONDITIONS: Diabetes Mellitus; Chronic Kidney Disease; Anemia
MeSH Terms: conditions — Diabetes Mellitus; Renal Insufficiency, Chronic; Anemia | interventions — Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Receive Darbepoetin alfa
  Interventions: Drug: Darbepoetin alfa
- 2 (No Intervention)

INTERVENTIONS:
Drug: Darbepoetin alfa — Starting dose of 20 microgram per week, to be titrated over a 3-month period until target hemoglobin level is reached (female: 11 g/dL and male: 12 g/dL). Route of administration is subcutaneous injection.
  Arms: 1

SUMMARY:
The purpose of this study is to examine the effect of partial correction of anemia with Darbepoetin alfa to a target of 11 g.dL (female) or 12 g/dL (male) on the reduction of cardiovascular morbidity and total mortality.

DETAILED DESCRIPTION:
Diabetes is the leading cause of end stage renal disease and cardiovascular disease with 60 percent of the global diabetic population coming from Asia. Growing evidence confirms the predictive role of chronic kidney disease (CKD) on cardiovascular morbidity and mortality. This is due to the constellation of conventional and non-conventional risk factors in patients who develop CKD, such as anemia, inflammation and abnormal bone metabolism. In this regard, anemia is a risk factor for cardiovascular disease and all-cause mortality in patients with CKD, patients with left ventricular dysfunction and in general population.

Effective erythropoiesis is dependent on the production of erythropoietin by the kidneys. Anemia is a common finding in patients with diabetes and up to 20% of diabetic patients are noted to have anemia. In a meta-analysis of community-based population studies, anemia interacts with CKD to increase the risk of coronary heart disease, stroke and all-cause mortality among patients with diabetes. Previous studies that examined the effect of erythropoietin therapy on anemic subjects with CKD did not find statistical difference in mortality rates between the treated and untreated groups. Possible explanations for the lack of benefits include higher level of blood pressure and increased blood viscosity leading to worsening of chronic congestive heart failure in the treated subjects. We hypothesize that partial correction of hemoglobin may be more appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged above 20 years old
* Patients with Type 1 or Type 2 diabetes mellitus
* Estimated glomerular filtration rate less than 59 mL/min/1.73m2
* Patients not on renal replacement therapy
* Hemoglobin level at baseline : women less than 9.5 g/dL (inclusive) and men less than 10.5 g/dL (inclusive)
* All patients should be on a stable dose of the following medications 4 weeks before enrolment :
* Aspirin 80mg daily unless contraindicated
* Statin to achieve stable and optimal LDL-cholesterol level
* Maximal tolerated dose of angiotensin-converting enzyme inhibitors or angiotensin receptor blockers
* Anti-hypertensive treatment to maintain blood pressure target of less than 130/80 mmHg or a level achieved without undue side effects
* Oral anti-diabetic drugs or insulin to maintain HbA1C less than 9.5%

Exclusion Criteria:

* Pregnancy, breast feeding or patient has plans of becoming pregnant during the study period
* Known non-diabetic renal disease
* Known cause of anemia not related to chronic kidney disease
* Presence of hemoglobinopathy
* History of pure red cell aplasia
* Known allergy to Darbepoetin alfa
* Severe liver impairment (>= 3x ULN of ALT)
* Poorly controlled hypertension, systolic BP >= 160mmHg or diastolic BP >= 100mmHg
* Significant cardiovascular disease within 3 months of enrolment including acute coronary syndrome, cardiac revascularization procedure, transient ischemic attack and cerebrovascular accident
* History of major gastrointestinal bleeding in the 5 years prior to consent
* Investigational drugs within 30 days of enrolment
* Any other medical conditions that is considered as unsuitable for the study by investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Composite cardiovascular endpoint of myocardial infarction, congestive heart failure, arrhythmia, stroke, transient ischemic attack, amputation or ulceration / necrosis of lower limb | 3 years
Death | 3 years

SECONDARY OUTCOMES:
Doubling of mean serum creatinine | 3 years
50% reduction in mean estimated glomerular filtration rate during baseline period as estimated by the abbreviated Modification of Diet in Renal Disease equation | 3 years
Estimated glomerular filtration rate less than 15 mL/min/1.73m-2 | 3 years
Change in fasting urinary albumin creatinine ratio | 3 years
Need for dialysis | 3 years
Number of hospital admissions, total number of days of hospital stay and attendance at the Accident and Emergency Department | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter CY Tong, MBChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, China